CLINICAL TRIAL: NCT06296316
Title: Real-Life Use of Transabdominal Restorelle® Meshes in Apical Prolapse Repair: an Observational Post-Market Clinical Study
Brief Title: Real-Life Use of Transabdominal Restorelle® Meshes in Apical Prolapse Repair
Acronym: REPAIR
Status: Terminated | Type: Observational
Why Stopped: From June 08, 2024, the study device was no longer marketed in France. Therefore, the sponsor decided to terminate the study prematurely.
Sponsor: Coloplast A/S (Industry)
Collaborators: International Clinical Trials Association (Other)
Responsible Party: Sponsor
Other Study IDs: IU022
Record Dates: First submitted 2023-11-24; First posted 2024-03-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Genital Prolapse
Keywords: Apical prolapse; Transabdominal mesh; Pelvic organ prolapse; Sacrocolpopexy; Sacrocervicopexy; Sacrohysteropexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Restorelle Polypropylene Mesh — The Coloplast Restorelle® Polypropylene Mesh is a Class III, implantable, permanent, non-absorbable, single use device indicated to restore female pelvic floor anatomy by providing anatomical support and suspension as a bridging material to support deficient fascia that resulted in descent of the female pelvic organs (pelvic organ prolapse).
  Restorelle mesh is a synthetic, macroporous mesh constructed of medical grade knitted, monofilament polypropylene.

SUMMARY:
The purpose of this study is to prospectively follow patients after a sacrocolpopexy with Restorelle® mesh for apical prolapse repair as part of routine care. It will help to describe the safety profile and to confirm the clinical benefits of Restorelle mesh for at least 5 to 8 years post-surgery.

DETAILED DESCRIPTION:
This study is a non-interventional, multicenter and post market clinical follow-up in adult women with apical prolapse under normal conditions of use (after a sacrocolpopexy with Restorelle mesh for apical prolapse repair as part of routine care). The patient will be followed for 1 year (or less) by the investigator as per local usual practice. At the same time, the patient will be followed via PRO (Patient Reported Outcomes) over a period of 5 to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Female patient of at least 18 years old
* Patient presenting apical pelvic organ prolapse and being eligible to surgical treatment
* Surgeon having decided to treat the patient with a Restorelle mesh as per its CE mark indication and IFU, before patient inclusion
* Patient having received appropriate information and counselling before mesh implantation
* Patient has been provided written informed consent

Exclusion Criteria:

* Patient currently pregnant or breastfeeding
* Patient being deprived of liberty by a judicial or administrative decision, or who is under a measure of legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients presenting with apical pelvic organ prolapse which is clinically indicated for a surgical treatment with Restorelle mesh
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
The incidence rate of a surgical reintervention related to Restorelle mesh use over at least the 5 first years of post-index procedure follow-up | up to 5 years

SECONDARY OUTCOMES:
Incidence rate of surgical reintervention related to Restorelle mesh use in patients | through study completion, at least 5 and up to 8 years
Number of patients who have only had surgical reintervention not related to Restorelle mesh use | through study completion, at least 5 and up to 8 years
Percentage of patients who have only had surgical reintervention not related to Restorelle mesh use | through study completion, at least 5 and up to 8 years
Number of patients who have had more than 1 surgical reintervention (unrelated to mesh use) | 5 years ; up to 8-year after index procedure
Percentage of patients who have had more than 1 surgical reintervention (unrelated to mesh use) | 5 years ; up to 8-year after index procedure
Description of patients who have had more than 1 surgical reintervention (unrelated to mesh use) | 5 years ; up to 8-year after index procedure
Patient impression of improvement of surgical reintervention assessed by the PGI-I-Reintervention | 6 months after surgical reintervention
  Patient Global Impression of Improvement (PGI-I) is a 7-point scale that provides a single global measure of condition improvement from 'very much better' to 'very much worse' after treatment. The surgery is defined as successful if the patient felt "very much better" or "much better". In case of reintervention, the patient will complete a PGI-I-Reintervention (same questionnaire as PGI-I) at 6 months after surgical reintervention.
Number of Adverse Device Effect | through study completion, at least 5 and up to 8 years
Percentage of Adverse Device Effect | through study completion, at least 5 and up to 8 years
Number of Restorelle mesh Device Deficiencies | through study completion, at least 5 and up to 8 years
Percentage of Restorelle mesh Device Deficiencies | through study completion, at least 5 and up to 8 years
Description of Restorelle mesh Device Deficiencies | through study completion, at least 5 and up to 8 years
  The description of identified Restorelle mesh Device Deficiencies and categorized according to the association or not with Adverse Device Effect (ADE) or Serious ADE
Monitoring of postoperative pain related to Restorelle mesh use using the modified TOMUS/PREM questionnaire | through study completion, at least 5 and up to 8 years
  Post-operative pain will be reported and evaluated by the patient using the modified TOMUS/PREM questionnaire through:
  * Location and Intensity VAS
  * Pain duration: acute or chronic (more than 6 months)
  * Treatment: types, drug name (if medication) and duration
  * Persistent pain, beyond 2 weeks, will be defined as having
    1. pain intensity ≥ 40 (VAS) at any of locations (lower abdomen, vagina, lower back and back of legs/buttocks) or during any activity or
    2. pain medication use.
Changes of prolapse symptoms | Pre-index procedure ; 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  The changes in the Pelvic Floor Disability Index (PFDI-20 questionnaire) total score and sub scores.
  Pelvic Floor Distress Inventory (PDFI-20) is comprised of 3 subscales for a total of 20 questions. Each question begins with a "yes" or "no" response. If "yes," the patient must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100 (with higher scores indicating more distress/dysfunction). The sum of the 3 scales are added together to get the PFDI-20 summary score, which ranges from 0 to 300.
Prolapse symptoms - number | 12 months ; 5 years
  The number of patients rating "yes" at "vaginal bulge" determined by the PFDI-20/POPDI-6 and requiring additional treatment for POP since index procedure
Prolapse symptoms - percentage | 12 months ; 5 years
  The percentage of patients rating "yes" at "vaginal bulge" determined by the PFDI-20/POPDI-6 and requiring additional treatment for POP since index procedure
Assessment of health related quality of life using the EQ-5D-5L questionnaire | Pre-index procedure ; 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  The changes in QoL total score using EQ-5D-5L and their evolution. The General Health Outcome Status questionnaire (EQ-5D-5L) consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions which are divided into 5 levels of perceived problems: from level 1 indicating no problem to level 5 indicating extreme problems. The patient indicates her health state in each of the 5 dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, from 'The best health you can imagine' to 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgment.
Assessment of health related quality of life using the PFIQ-7 questionnaire | Pre-index procedure ; 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  The changes in QoL total score using the Pelvic Floor Impact Questionnaire (PFIQ-7) and their evolution.
  Pelvic Floor Impact Questionnaire (PFIQ-7) consists of 7 questions. The responses for each question range from "not at all" (0) to "quite a bit" (3). To get scale scores, the mean of each of the 3 scales is individually calculated, which ranges from 0-3, this number is then multiplied by 100 and then divided by 3. The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life.
Assessment of the sexual functioning by the PISQ-IR questionnaire | Pre-index procedure ; 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA revised (PISQ-IR): is composed of 20 items including the scales for arousal & orgasm, partner related, condition specific, global quality, condition impact and desire. The number of cases for each scale that can be scored. The mean and standard deviation are provided for each scale.
Assessment of the sexual functioning by the changes in dyspareunia status of patients who are sexually active. | Pre-index procedure ; 12 months
Number of patients defining success via patient global impression of improvement (PGI-I) scale | 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  Patient Global Impression of Improvement (PGI-I) is a 7-point scale that provides a single global measure of condition improvement from 'very much better' to 'very much worse' after treatment. The surgery is defined as successful if the patient felt "very much better" or "much better".
Percentage of patients defining success via patient global impression of improvement (PGI-I) scale | 2 months ;12 months ; Every year (at least 5 and up to 8 years)
  Patient Global Impression of Improvement (PGI-I) is a 7-point scale that provides a single global measure of condition improvement from 'very much better' to 'very much worse' after treatment. The surgery is defined as successful if the patient felt "very much better" or "much better".
Number of patients satisfied after the index procedure as assessed by the Surgical Satisfaction Questionnaire (SSQ-8). | 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  Surgical Satisfaction Questionnaire (SSQ-8): is a validated questionnaire used to measure patient satisfaction following a surgery to correct prolapse and/or incontinence. Answers of the SSQ questions consisted of a 5-point scale ranging from "very satisfied" to "very unsatisfied" or from "yes" to "never". Patients' satisfaction is defined if answers correspond with "very satisfied" and "satisfied" or "yes" and "may be".
Percentage of patients satisfied after the index procedure as assessed by the Surgical Satisfaction Questionnaire (SSQ-8) | 2 months ; 12 months ; Every year (at least 5 and up to 8 years)
  Surgical Satisfaction Questionnaire (SSQ-8): is a validated questionnaire used to measure patient satisfaction following a surgery to correct prolapse and/or incontinence. Answers of the SSQ questions consisted of a 5-point scale ranging from "very satisfied" to "very unsatisfied" or from "yes" to "never". Patients' satisfaction is defined if answers correspond with "very satisfied" and "satisfied" or "yes" and "may be".

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ferry, Dr, Principal Investigator — CH La Rochelle, France
Locations (6):
- France (6):
  - Polyclinique de la Baie, Avranches, Choisir Une Région
  - CHU Pellegrin, Bordeaux
  - CH La Rochelle, La Rochelle
  - Clinique Bon Secours, Le Puy-en-Velay
  - Institut Mutualiste Montsouris, Paris
  - CH de Saintonge, Saintes

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available